CLINICAL TRIAL: NCT07402395
Title: Efficacy and Safety of BtH Intimate 2.0% (Injectable Cross-Linked Hyaluronic Acid) in the Volumization and Aesthetic Rejuvenation of the Female Vulvovaginal Area: A Prospective Clinical Investigation
Brief Title: Clinical Study on the Safety and Efficacy of an Injectable Hyaluronic Acid for Improving the Aesthetic Rejuvenation of the Vulvovaginal Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Dr. Goya Análisis, SL. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BtHCi-PIC01-2024
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Vulvar Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BtHIntimate® Injectable Hyaluronic Acid Treatment (Experimental): Participants in this single-arm study will receive a single intradermal infiltration of BtH Intimate 2.0% intended to restore volume and improve the aesthetic appearance, hydration, and firmness of the vulvovaginal area.
  Interventions: Device: BtHIntimate® Injectable Hyaluronic Acid Treatment

INTERVENTIONS:
Device: BtHIntimate® Injectable Hyaluronic Acid Treatment — BtHIntimate 2.0% is administered to the labia majora and/or mons pubis according to individual clinical needs. An optional touch-up may be performed at the 4-week follow-up visit if deemed necessary by the investigator. All participants are followed for 6 months, during which aesthetic outcomes, tissue hydration, patient-reported symptoms, sexual function, satisfaction, and safety events are evaluated.

SUMMARY:
This prospective, single-center, before-after study evalutated BtH Intimate 2.0%, a cross-linked hyaluronic acid injectable used to restore volume and improve the aesthetic appearance and hydration of the vulvovaginal area in adult women. Forty participants with mild to moderate vulvar atrophy or genital aging signs received a single treatment, with an optional touch-up at 4 weeks, and were followed for six months. The primary objectives were to measure global aesthetic improvement using the GAIS scale and to assess safety through the recording of serious adverse events. Secondary measures included patient satisfaction, sexual function (FSFI), symptom improvement (VAS), tissue hydration, and overall patient-reported benefit. Expected risks were mild and transient, consistent with HA fillers, while the intervention aimed to enhance comfort, appearance, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥18 years).
* Women with mild or moderate vulvar atrophy, including deflation or vulvar ptosis, or with visible signs of genital aging, or women seeking aesthetic improvement of the vulvovaginal area, including peri-menopausal or women with genitourinary syndrome of menopause (GSM).
* Ability and willingness to comply with all study visits and procedures.
* Sufficient predisposition and capacity, in the investigator's judgment, to complete study questionnaires.
* For women of childbearing potential: negative pregnancy test and agreement to use reliable contraception during the study (hormonal contraception, IUD/IUS, condoms, diaphragm with spermicide, vasectomized partner, or true abstinence).

Exclusion Criteria:

* Allergy or hypersensitivity to any component of BtH Intimate 2.0%.
* Pregnancy or planned pregnancy, or breastfeeding.
* Active infection or pathology in the area to be treated.
* Presence of bacterial, fungal, or viral infection in or near the vulvovaginal region, or current treatment for such conditions.
* Known tendency to develop hypertrophic scars or keloids.
* Signs of inflammation in or near the treatment area, or receiving treatment for inflammation.
* History of any vulvovaginal rejuvenation procedure within the last 6 months or during the study (e.g., laser, radiofrequency, electrotherapy, dermal fillers, PRP, etc.).
* Unrealistic or disproportionate expectations regarding treatment outcomes.
* Incorrectly selected participants (those found retrospectively to fail inclusion or meet exclusion criteria) will be replaced.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Global Aesthetic Improvement (GAIS) | Baseline to 12 weeks and 24 weeks
  Aesthetic improvement of the vulvovaginal area assessed by the investigator using the 5-point Global Aesthetic Improvement Scale (GAIS: "very much improved," "much improved," "improved," "no change," "worse"). Clinical relevance is defined as ≥60% of participants rated as "Improved" or better at week 12 or 24.
Incidence of Serious Adverse Events (SAEs) | 6 months
  Number, frequency, severity, and relationship of all serious adverse events recorded according to EU MDR definitions (death, life-threatening events, hospitalization, permanent impairment, or fetal harm).

SECONDARY OUTCOMES:
Patient Satisfaction (Likert Scale) | Immediatly post-treatment, at 4 weeks, at 12 weeks and at 24 weeks
  A 5 point Likert Scale (Very satisfied, Satisfied, Slightly satisfied, indifferent and unsatisfied). The percentage of very satisfied, satisfied and slightly satisfied answers was taken into account.
Investigator-Rated Aesthetic Parameters with a Visual Analogue Scale (VAS) | Baseline, 4 weeks, 12 weeks, 24 weeks
  Clinical assessment of improvement in aesthetic parameters using a visual analogue scale (VAS 0-10): volume, hydration, elasticity, hyperpigmentation, and firmness. Improvement will be calculated as the change in points from baseline.
Female Sexual Function Index (FSFI) | Baseline, 4 weeks, 12 weeks, 24 weeks
  The FSFI consists of 19 multiple-choice questions coded from 0.0 to 5.0. Each score has a specific meaning depending on the item. The scale includes six sexual domains. The maximum score for each domain is 6.0, obtained by summing the item responses and multiplying by a correction factor. The total composite sexual function score is the sum of all domain scores and ranges from 2.0 (not sexually active and no desire) to 36.0. Improvement will be calculated as the change in points from baseline.
Vulvovaginal Symptoms (VAS) | Baseline, 4 weeks, 12 weeks, 24 weeks
  Vulvovaginal symptoms assessed using a 0-10 visual analogue scale (VAS). The following symptoms are evaluated: itching, friction or rubbing associated with atrophy, dryness, pain, sensitivity, tingling, and dyspareunia. Improvement will be calculated as the change in points from baseline.
PGI-I (Patient Global Impression of Improvement) | Time Frame: 4 weeks, 12 weeks, 24 weekS
  Patient's global impression of improvement using 7-point PGI-I scale (1 = "very much improved" to 7 = "very much worse"). Responders are scores 1 (Very much improved), 2 (Much improved) and 3 (Improved).
Hydration of Vulvar Tissue (Corneometer®) | Baseline, 4 weeks, 12 weeks, 24 weeks
  Hydration of the treated area measured using a Corneometer® biometric probe. Improvement will be calculated relative to baseline values."
Non-Serious Adverse Events (AEs) | 6 months
  Frequency, severity, duration, and investigator-determined causality of all non-serious adverse events (e.g., erythema, swelling, bruising, palpable nodules).
Future Use Questionnaire | 24 weeks
  Participant-reported acceptance and willingness to use the product again or recommend it, including purchase intention and perceived effectiveness.
Usability Assessment (Investigator) | 24 weeks
  Investigator evaluation of device usability, including syringe handling, injection force, ergonomics, packaging, and product flow through the cannula.

CONTACTS AND LOCATIONS:
Locations (1):
- Complutense Medical Center (Virtus Group), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No